CLINICAL TRIAL: NCT00898170
Title: Effect of Myoma Removal on Blood Pressure and Erythropoetin Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: javad Kojuri, shiraz university of medical sciences
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 88-2505
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Myoma; Hypertension
Keywords: myoma; hypertension; erythropoetin; blood pressure; erythropoetin level
MeSH Terms: conditions — Myoma; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- myoma, with or without hypertension (Experimental): those with myoma with or without hypertension in holter monitoring
  Interventions: Procedure: myoma removal

INTERVENTIONS:
Procedure: myoma removal — surgical removal of myoma by hysterectomy

SUMMARY:
The effect of myoma removal was studied on 28 patients with hypertension and myoma by holter monitoring and erythropoetin level check.

DETAILED DESCRIPTION:
Background:

Myoma is the most common gynecoid tumor and produces many vasoactive substances, which may be a cause for secondary hypertension. Early reports suggested the association of myoma and hypertension. We studied the effect of myoma removal on hypertension and erythropoietin level to evaluate this hypothesis.

Patients & Methods:

In this single centered prospective cohort study, in twenty eight patients who were candidates for myomectomy due to myoma, 24 hour holter monitoring of blood pressure and serum erythropoietin were checked before and 6 weeks after hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* candidate for myoma removal by hysterectomy
* operable
* hysterectomy is indicated

Exclusion Criteria:

* patient refusal
* inoperable patients
* other secondary cases of hypertension

Ages: 22 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
24 hour holter monitoring of blood pressure | 6 weeks

SECONDARY OUTCOMES:
erythropoetin level | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: javad kojuri, M.D., Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Cardiology Ward Shiraz University of Medical Sciences, Shiraz, Fars, Iran